CLINICAL TRIAL: NCT02905643
Title: The Use of Peak Height and Percentage Signal Recovery for Evaluation and Determination of Pseudoprogression in Glioblastoma Patients
Brief Title: Discerning Pseudoprogression vs True Tumor Growth in GBMs
Status: Terminated | Type: Observational
Why Stopped: Investigator left institution
Sponsor: Ascension Health (Industry)
Responsible Party: Sponsor
Other Study IDs: R20150109
Record Dates: First submitted 2016-09-08; First posted 2016-09-19 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma
Keywords: Pseudoprogression; Brain Cancer
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study subjects: Patients who have or might have a brain tumor which may be a glioblastoma.
  Interventions: Other: Study subjects

INTERVENTIONS:
Other: Study subjects — This study does not include an intervention it is only observational.

SUMMARY:
One-third of all primary brain tumors are astrocytomas, the most common type of glioma. Grade 4 astrocytomas, more commonly known as glioblastomas (GBMs), represent about 50% of all gliomas (annual incidence of over 3 per 100,000) and are associated with high mortality rates and median patient survival of just 12-15 months post-diagnosis. Treatment response is assessed by measuring post-treatment tumor size on contrast-enhanced magnetic resonance images (MRI). However, radiation and chemotherapy cause inflammatory and necrotic changes which, like actual tumor progression itself, demonstrate contrast enhancement on the first post-treatment MRI scan. This enhancement eventually subsides (typically within 6 months of treatment) and is known as pseudoprogression (PsP). Currently, there is no gold standard noninvasive tool for distinguishing between pseudoprogression and progressive disease. Dynamic susceptibility-weighted contrast-enhanced perfusion MRI (DSC perfusion MRI) permits measurement of hemodynamic imaging variables. Previous literature reports attempted to use some or all of these metrics to assess their utility in distinguishing PsP from true cancer progression. These studies showed mixed results, likely due to a number of factors, including poor statistical power, poorly defined PsP, analysis of multiple cancer grades and types, and varied analysis methodologies. The investigators aim to address these issues in this study.

DETAILED DESCRIPTION:
See BRIEF SUMMARY section

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older.
* Participants must be able to read and comprehend the English language.
* In agreement with the care providing physician, participants must be willing to have surgery to remove possible brain tumor.
* Participants must have a MRI scan within 24 hours after the tumor is removed (if a tumor is confirmed).
* Participants must have the tumor analyzed by the laboratory and pathology departments and receive the diagnosis of glioblastoma.
* Participants must be willing to follow the Stupp treatment protocol (this treatment plan and its' procedures are considered the standard for treating glioblastoma). (The Stupp protocol is the name of the radiation and chemotherapy plan that has been found to help in many cases of glioblastoma.)
* Participants must be willing to follow any additional study procedures (including having all follow-up MRIs performed at St. Vincent 86th St).

Exclusion Criteria:

* Participants are less than 18 years of age.
* Participants have had surgery for your brain tumor and NOT received the diagnosis of glioblastoma
* Participants and care providing physician have decided NOT to follow the Stupp protocol (treatment plan) for glioblastoma treatment. (Deviations or interruptions are allowed if clinically indicated)
* Participants are not having a MRI scan within 24 hours after brain tumor surgery.
* Participants are not willing to follow the study procedures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have or might have a brain tumor which may be a glioblastoma.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Imaging parameter utility for pseudoprogression vs. true tumor growth | Up to 24 months
  The primary outcome of this study is to assess the utility of peak height, peak signal recovery, apparent diffusion coefficient, and cerebral blood volume (and their relative values) in determining, positive predictive values (PPV), negative predictive values (NPV), and likelihood ratios (LR) for identifying pseudo progression versus true tumor growth.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Beltz, MD, Principal Investigator — Northwest Radiology Network, Inc

IPD SHARING:
Plan to Share IPD: No